CLINICAL TRIAL: NCT01017965
Title: Impact of Objective Sleep Duration on Blood Glucose Control in Type 1 Diabetes Adult Patients
Acronym: DIAPASOM2
Status: Terminated | Type: Observational
Why Stopped: intermediary analysis was performed and significant results were found for the main objective
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 0917; 2009-A00816-51 (Registry Identifier: ID CRB)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Pressure Monitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A sample of serum will be retained in order to compare indicators of inflammation with sleep duration and diabetes complications
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Actimeter + blood pressure monitoring — Patients will receive an actimeter that they will wear for 3 days and an ambulatory blood pressure monitoring device that they will keep for 24 hours.
  Other Names: Actiwatch-16, Mini-Mitter Inc, Bend,Oregon; SPACELABS 90207

SUMMARY:
The objective of this study is to assess the impact of objective sleep duration on blood glucose control in type 1 diabetes adult patients.

This study will also evaluate the impact of objective sleep duration on blood pressure over a 24-hour period and the impact of objective sleep duration on quality of life.

Last, it will investigate the influence of objective physical activity duration on blood glucose control, blood pressure and quality of life.

DETAILED DESCRIPTION:
The objective of this study is to assess the impact of objective sleep duration on blood glucose control in type 1 diabetes adult patients.

This study will also evaluate the impact of objective sleep duration on blood pressure over a 24-hour period and the impact of objective sleep duration on quality of life.

Last, it will investigate the influence of objective physical activity duration on blood glucose control, blood pressure and quality of life.

This study will enrol ambulatory patients only. On day 0, patients receive an actimeter and an ambulatory blood pressure monitoring device. The actimeter measures activity and sleep duration. The patient keeps the actimeter for 3 consecutive days and the blood pressure monitoring device for 24 hours. A blood sample is also collected.

Patients will be divided into 2 groups, based on objective sleep duration: 'short-sleepers' and 'long-sleepers'. The threshold will be the median of the total population. HbA1c will be compared between the 2 groups with a Student test or a Mann-Whitney test, depending on the normality of distribution.

A model of multiple linear regression will be created. HbA1c will be entered as dependant variable and objective sleep duration as independent variable

Patients will be divided into 2 groups, based on objective activity duration: 'low-activity' and 'high-activity'. The threshold will be the median of the total population. HbA1c, blood pressure, quality of life, biological results and general characteristics will be compared between the 2 groups with a Student test or a Mann-Whitney test, depending on the normality of distribution. Qualitative variables will be studied with a chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to Social Security
* Written consent to participate to the study
* Ambulatory medical follow-up
* Patient with type 1 diabetes, defined by the criteria of the American Diabetes Association in 1997, stable (no ketoacidosis episode or hypoglycaemia with loss of consciousness requiring the intervention of a third person, during the previous month)

Exclusion Criteria:

* Underage patient, major patient under guardianship or protected by the Law
* Pregnant, parturient or breastfeeding woman
* Person with no freedom (prisoner), person hospitalized without consent and not protected by the Law
* Non-stabilized diabetes with at least one ketoacidosis episode or hypoglycaemia with loss of consciousness requiring the intervention of a third person, during the previous month.
* Bedridden person or person with mobility impairment.
* Patient already hospitalized at enrolment time
* Patient whose physical or psychological health could interfere with obtention of informed consent and compliance to the protocol (especially answers to the questionnaires)
* Terminally-ill patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll type 1 diabetes patients who come for a consultation in Grenoble University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
HbA1c in % | Day 0 or Day 3

SECONDARY OUTCOMES:
Objective sleep duration in minutes | Day 0 to Day 3
Blood pressure in cm Hg | Day 0, 24 hours
Quality of life assessed through questionnaire | Day 0 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Benhamou, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Service de Diabétologie du Pr Halimi, CHU, Grenoble, France

REFERENCES:
- [Derived] Borel AL, Pepin JL, Nasse L, Baguet JP, Netter S, Benhamou PY. Short sleep duration measured by wrist actimetry is associated with deteriorated glycemic control in type 1 diabetes. Diabetes Care. 2013 Oct;36(10):2902-8. doi: 10.2337/dc12-2038. Epub 2013 May 28. PMID 23715755